CLINICAL TRIAL: NCT03610009
Title: Manual Versus Automated Measurements of Ovarian Follicle Diameter in High Responding Patients With GnRH Agonist Triggering of Final Oocyte Maturation
Brief Title: 2D Versus SonoAVC Scanning in High Responders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SonoAVC
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Follicle development in women undergoing IVF will be monitored either by conventional 2D ultrasound or SonoAVC.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Women (patients), clinician performing oocyte retrieval and clinical embryologist will be blinded to the method used for monitoring follicle development
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2D ultrasound (Active Comparator): Two-dimensional (2D) ultrasound is used to identify number and size of ovarian follicles, to select optimal day for triggering final oocyte maturation.
  Interventions: Device: 2D ultrasound
- SonoAVC (Active Comparator): SonoAVC is used to identify number and size of ovarian follicles, to select optimal day for triggering final oocyte maturation.
  Interventions: Device: SonoAVC

INTERVENTIONS:
Device: 2D ultrasound — The timing of final follicle maturation and oocyte retrieval based on follicle tracking with use of conventional two-dimensional (2D) ultrasound.
  Arms: 2D ultrasound
Device: SonoAVC — The timing of final follicle maturation and oocyte retrieval based on follicle tracking with use of SonoAVC.
  Arms: SonoAVC

SUMMARY:
Accurate follicular monitoring of Controlled Ovarian Stimulation by transvaginal ultrasound is considered important for the success of human in vitro fertilization (IVF). The aim of this study is to evaluate the effect of timing oocyte maturation and egg collection on the basis of follicular measurements made automatically with Sono Automated Volume Calculation (SonoAVC) against those made with conventional 2D ultrasound in relation to the number of mature oocytes collected.

This study will take place in women undergoing IVF who are high responders (>=14 follicles>=11mm) and hence at risk for developing ovarian hyperstimulation syndrome (OHSS), treated with a GnRH antagonist protocol and administered GnRH agonist to trigger final oocyte maturation.

DETAILED DESCRIPTION:
Accurate follicular monitoring of Controlled Ovarian Stimulation by transvaginal ultrasound is considered important for the success of human in vitro fertilization (IVF). Accurate assessment of the size of follicles is important for the timing of oocyte maturation and subsequent oocyte retrieval.

Serial assessment of follicle number and size is used routinely to assess the response to ovarian stimulation during assisted reproduction treatment (ART). Two-dimensional (2D) ultrasound is used to identify and scroll through each ovary while the observer quantifies the number of follicles present. An objective assessment of the size of the larger follicles, commonly those measuring >10 mm, is then made through a series of 2D measurements of their perceived mean diameter.

Sono Automated Volume Calculation (SonoAVC; GE Medical Systems) is a new software program that can be applied to datasets acquired with use of threedimensional (3D) ultrasound. It individually identifies and quantifies the size of any hypoechoic region within these 3D datasets, providing an automatic estimation of their absolute dimensions and volume. SonoAVC is an ideal and, potentially, a clinically important tool for the assessment and measurement of follicles during controlled ovarian stimulation because each hypoechoic area is individually color coded, thereby eliminating the possibility of measuring the same follicle more than once.

In women with high ovarian response to gonadotrophin stimulation, the accurate measurement of the number and size of follicles present in hyperstimulated ovaries is a challenge for clinicians and ultrasonographers.

The aim of this study is to evaluate the effect of timing final oocyte maturation trigger and egg collection on the basis of follicular measurements made automatically with SonoAVC against those made with conventional 2D ultrasound in relation to the number of mature oocytes collected. This study will include women undergoing ART who are high responders (presence of =>14 follicles>=11mm) and hence at risk for developing ovarian hyperstimulation syndrome (OHSS), treated with a GnRH antagonist protocol and are administered GnRH agonist to trigger final oocyte maturation. All resulting embryos (blastocysts) will be cryopreserved and transferred in a subsequent frozen cycle.

ELIGIBILITY:
Inclusion Criteria:

* AMH >= 3ng/ml
* at least 14 follicles =>11 mm diameter on final day of stimulation
* undergoing GnRH antagonist protocol
* administered GnRH agonist to trigger final oocyte maturation

Exclusion Criteria:

* poor responders
* hCG injection to trigger final oocyte maturation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of mature oocytes | Day of oocyte retrieval
  The number of mature (metaphase-II) oocytes retrieved

SECONDARY OUTCOMES:
Number of oocytes retrieved | Day of oocyte retrieval
  Total number of oocytes retrieved
Oocyte maturation rate | Day of oocyte retrieval
  Percentage of mature oocytes/total number of oocytes
Oocyte retrieval rate | Day of oocyte retrieval
  Percentage of oocyte retrieved/number of follicles aspirated
Number of fertilised oocytes | 1 day post oocyte retrieval
  Number of fertilised oocytes displaying 2 pronuclei and 2 polar bodies
Fertilisation rate | 1 day post oocyte retrieval
  Percentage fertilised oocytes/oocytes inseminated
Number of blastocysts | 5 days post oocyte retrieval
  Number of embryos reaching the blastocyst stage
Days of stimulation | 10-15 days after menses
  Number of days recFSH is administered
Total dose of recFSH | 10-15 days after menses
  Total dose of recFSH administered during the ovarian stimulation period

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon Lainas, PhD, Study Director — Eugonia
Locations (1):
- Eugonia Unit of Assisted Reproduction, Athens, Greece

REFERENCES:
- [Background] Raine-Fenning N, Deb S, Jayaprakasan K, Clewes J, Hopkisson J, Campbell B. Timing of oocyte maturation and egg collection during controlled ovarian stimulation: a randomized controlled trial evaluating manual and automated measurements of follicle diameter. Fertil Steril. 2010 Jun;94(1):184-8. doi: 10.1016/j.fertnstert.2009.02.063. Epub 2009 Apr 1. PMID 19342014
- [Background] Lamazou F, Arbo E, Salama S, Grynberg M, Frydman R, Fanchin R. Reliability of automated volumetric measurement of multiple growing follicles in controlled ovarian hyperstimulation. Fertil Steril. 2010 Nov;94(6):2172-6. doi: 10.1016/j.fertnstert.2010.01.062. Epub 2010 Mar 12. PMID 20226448
- [Background] Salama S, Arbo E, Lamazou F, Levailllant JM, Frydman R, Fanchin R. Reproducibility and reliability of automated volumetric measurement of single preovulatory follicles using SonoAVC. Fertil Steril. 2010 Apr;93(6):2069-73. doi: 10.1016/j.fertnstert.2008.12.115. Epub 2009 Apr 1. PMID 19342038
- [Background] Ata B, Seyhan A, Reinblatt SL, Shalom-Paz E, Krishnamurthy S, Tan SL. Comparison of automated and manual follicle monitoring in an unrestricted population of 100 women undergoing controlled ovarian stimulation for IVF. Hum Reprod. 2011 Jan;26(1):127-33. doi: 10.1093/humrep/deq320. Epub 2010 Nov 26. PMID 21112951
- [Background] Rodriguez-Fuentes A, Hernandez J, Garcia-Guzman R, Chinea E, Iaconianni L, Palumbo A. Prospective evaluation of automated follicle monitoring in 58 in vitro fertilization cycles: follicular volume as a new indicator of oocyte maturity. Fertil Steril. 2010 Feb;93(2):616-20. doi: 10.1016/j.fertnstert.2009.02.058. Epub 2009 Apr 18. PMID 19376513
- [Background] Revelli A, Martiny G, Delle Piane L, Benedetto C, Rinaudo P, Tur-Kaspa I. A critical review of bi-dimensional and three-dimensional ultrasound techniques to monitor follicle growth: do they help improving IVF outcome? Reprod Biol Endocrinol. 2014 Nov 24;12:107. doi: 10.1186/1477-7827-12-107. PMID 25420733
- [Background] Deb S, Campbell BK, Clewes JS, Raine-Fenning NJ. Quantitative analysis of antral follicle number and size: a comparison of two-dimensional and automated three-dimensional ultrasound techniques. Ultrasound Obstet Gynecol. 2010 Mar;35(3):354-60. doi: 10.1002/uog.7505. PMID 20069654
- [Background] Deutch TD, Joergner I, Matson DO, Oehninger S, Bocca S, Hoenigmann D, Abuhamad A. Automated assessment of ovarian follicles using a novel three-dimensional ultrasound software. Fertil Steril. 2009 Nov;92(5):1562-8. doi: 10.1016/j.fertnstert.2008.08.102. Epub 2008 Oct 19. PMID 18937942
- [Background] Vandekerckhove F, Bracke V, De Sutter P. The Value of Automated Follicle Volume Measurements in IVF/ICSI. Front Surg. 2014 May 28;1:18. doi: 10.3389/fsurg.2014.00018. eCollection 2014. PMID 25593942
- [Background] Pan P, Chen X, Li Y, Zhang Q, Zhao X, Bodombossou-Djobo MM, Yang D. Comparison of manual and automated measurements of monodominant follicle diameter with different follicle size in infertile patients. PLoS One. 2013 Oct 10;8(10):e77095. doi: 10.1371/journal.pone.0077095. eCollection 2013. PMID 24130840
- [Background] Raine-Fenning N, Jayaprakasan K, Chamberlain S, Devlin L, Priddle H, Johnson I. Automated measurements of follicle diameter: a chance to standardize? Fertil Steril. 2009 Apr;91(4 Suppl):1469-72. doi: 10.1016/j.fertnstert.2008.07.1719. Epub 2008 Oct 18. PMID 18930205
- [Background] Raine-Fenning N, Jayaprakasan K, Clewes J, Joergner I, Bonaki SD, Chamberlain S, Devlin L, Priddle H, Johnson I. SonoAVC: a novel method of automatic volume calculation. Ultrasound Obstet Gynecol. 2008 Jun;31(6):691-6. doi: 10.1002/uog.5359. PMID 18484679
- [Background] Broekmans FJ, de Ziegler D, Howles CM, Gougeon A, Trew G, Olivennes F. The antral follicle count: practical recommendations for better standardization. Fertil Steril. 2010 Aug;94(3):1044-51. doi: 10.1016/j.fertnstert.2009.04.040. Epub 2009 Jul 8. PMID 19589513
- [Background] Soldevila PN, Carreras O, Tur R, Coroleu B, Barri PN. Sonographic assessment of ovarian reserve. Its correlation with outcome of in vitro fertilization cycles. Gynecol Endocrinol. 2007 Apr;23(4):206-12. doi: 10.1080/09513590701253776. PMID 17505940